CLINICAL TRIAL: NCT00007657
Title: CSP #424 - Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation
Brief Title: Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Medical Research Council of Canada (Other); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); GE Healthcare (Industry); Bristol-Myers Squibb (Industry); Astellas Pharma Inc (Industry); AstraZeneca (Industry); Sanofi (Industry); Datascope Corp. (Industry); First Horizon (Unknown); Kos (Unknown); Key Pharmaceuticals (Industry); Integrated Therapeutics Group (Industry); Hoest-Marion-Roussel (Unknown)
Responsible Party: Boden, William - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 424
Record Dates: First submitted 2000-12-29; First posted 2001-01-04 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Myocardial Ischemia
Keywords: PCI plus intensive medical therapy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Percutaneous Coronary Intervention (PCI) plus intensive medical therapy
  Interventions: Procedure: Intensive medical therapy; Procedure: Percutaneous Coronary Intervention (PCI) plus intensive medical therapy
- 2 (Active Comparator): Intensive medical therapy
  Interventions: Procedure: Intensive medical therapy

INTERVENTIONS:
Procedure: Intensive medical therapy
Procedure: Percutaneous Coronary Intervention (PCI) plus intensive medical therapy
  Arms: 1

SUMMARY:
PCI (optimal catheter-based coronary revascularization) + intensive medical therapy is superior to intensive medical therapy alone using the combined endpoint of all-cause mortality or nonfatal MI.

DETAILED DESCRIPTION:
Primary Hypothesis: The strategy of PCI plus intensive medical therapy will be superior to intensive medical therapy alone in reducing all cause mortality or nonfatal MI in patients with documented myocardial ischemia who meet an AHA task force Class I indication for PCI.

Secondary Hypotheses: Resource utilization and QOL comparisons and hospitalization for acute coronary syndromes will be superior in PCI plus medical therapy compared to medical therapy alone.

Primary Outcomes: All cause mortality, nonfatal MI.

Interventions: All patients will be treated with intensive medical therapy. In addition half of them will receive percutaneous coronary intervention (PCI).

Study Abstract: The COURAGE Trial is a large-scale, multicenter, randomized controlled trial comparing medical therapy and PCI plus medical therapy that is powered for "hard" clinical endpoints. Patients eligible for inclusion in COURAGE will comprise all but very high-risk subjects, and will include those with chronic angina pectoris (Canadian Cardiovascular Society [CCS] Class I-III), recent uncomplicated MI, and asymptomatic (or "silent") myocardial ischemia. Patients may have single- or multi-vessel coronary artery disease and may have had prior bypass graft surgery or PCI. We project cumulative 3-year event rates of 16.4% and 21%, respectively, which yields an absolute difference of 4.6% or relative difference of 22%. With a minimum duration of follow-up of 2 1/2 years, a maximum of 7 years, using a two-sided test of significance at the 0.05 level, and assuming a 3% crossover rate then 2% then 1% each for 2 years from meds to PCI, and annual loss to follow-up rate of 1% these event rates indicate that a sample size of 2,270 will be needed to test the hypothesis with 85% power. Fifteen VA, 19 U.S. non-VA, and 16 Canadian sites enrolled in the study. The planned study duration was 7 years, with 4 1/2 years of patient intake and 2 1/2 - 7 years of follow-up. Study operations began in January 1999 and enrollment began in June 1999. The Data and Safety Monitoring Board approved reducing the sample size to 2,270 subjects based on increasing the length of randomization and follow-up and updating the definition of MI to include biomarker positive (troponin) ACS. Enrollment is complete with 2,287 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in COURAGE will comprise all but very high-risk subjects, and will include those with chronic angina pectoris (Canadian Cardiovascular Society [CCS] Class I-III), uncomplicated MI, cooled down ACS, and asymptomatic (or "silent") myocardial ischemia.
* Patients may have single- or multi-vessel coronary artery disease and may have had prior bypass graft surgery or PCI.

It is important to emphasize that as many types of CAD patients as possible--reflecting the spectrum of patients encountered in contemporary clinical practice--will be enrolled in COURAGE.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3260 (Estimated)
Dates: Start 1998-12; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E. Boden, Study Chair — VA South Texas Health Care System, San Antonio
Locations (48):
- United States (34):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - Southern CA Kaiser Permanente Medical Group, Los Angeles, California
  - VA Northern California HCS, Sacramento, California
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Systems-Newark, DE, Newark, Delaware
  - MIMA Century Research Associates - Melbourne, FL, Melbourne, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - Mayo Clinic Rochester - Rochester, MN, Rochester, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, St Louis, St Louis, Missouri
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - New York Harbor HCS, New York, New York
  - University of Rochester Strong Memorial Hospital, Rochester, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Portland, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA Medical Center, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
- Canada (14):
  - Foothills Hospital - Calgary, Alberta - Can, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St Paul's Hospital, Vancouver - British Columbia, Vancouver, British Columbia
  - St. John Regional Hospital Facility, Saint John, New Brunswick
  - Queen Elizabeth Ii Hsc, Halifax, Nova Scotia - Can, Halifax, Nova Scotia
  - Sudbury Regional Hospital - Sudbury, Ontario, Greater Sudbury, Ontario
  - Hamilton General Hospital - Hamilton, Ont - Can, Hamilton, Ontario
  - London Health Sciences Ctr - London, Ont - Can, London, Ontario
  - Trillium Health Care, Mississauga, Ontario
  - Sunnybrook HSC - Toronto, Ontario, Toronto, Ontario
  - St. Michael'S Hospital, Toronto, Ontario - Can, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute - Montreal, Quebec - Can, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Mancini GBJ, Maron DJ, Hartigan PM, Spertus JA, Kostuk WJ, Berman DS, Teo KK, Weintraub WS, Boden WE; COURAGE Trial Research Group. Lifestyle, Glycosylated Hemoglobin A1c, and Survival Among Patients With Stable Ischemic Heart Disease and Diabetes. J Am Coll Cardiol. 2019 Apr 30;73(16):2049-2058. doi: 10.1016/j.jacc.2018.11.067. PMID 31023428
- [Derived] Weintraub WS, Hartigan PM, Mancini GBJ, Teo KK, Maron DJ, Spertus JA, Chaitman BR, Shaw LJ, Berman D, Boden WE. Effect of Coronary Anatomy and Myocardial Ischemia on Long-Term Survival in Patients with Stable Ischemic Heart Disease. Circ Cardiovasc Qual Outcomes. 2019 Feb;12(2):e005079. doi: 10.1161/CIRCOUTCOMES.118.005079. PMID 30773025
- [Derived] Maron DJ, Mancini GBJ, Hartigan PM, Spertus JA, Sedlis SP, Kostuk WJ, Berman DS, Teo KK, Weintraub WS, Boden WE; COURAGE Trial Group. Healthy Behavior, Risk Factor Control, and Survival in the COURAGE Trial. J Am Coll Cardiol. 2018 Nov 6;72(19):2297-2305. doi: 10.1016/j.jacc.2018.08.2163. PMID 30384885
- [Derived] Zhang Z, Jones P, Weintraub WS, Mancini GBJ, Sedlis S, Maron DJ, Teo K, Hartigan P, Kostuk W, Berman D, Boden WE, Spertus JA. Predicting the Benefits of Percutaneous Coronary Intervention on 1-Year Angina and Quality of Life in Stable Ischemic Heart Disease: Risk Models From the COURAGE Trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation). Circ Cardiovasc Qual Outcomes. 2018 May;11(5):e003971. doi: 10.1161/CIRCOUTCOMES.117.003971. PMID 29752388
- [Derived] Sedlis SP, Hartigan PM, Teo KK, Maron DJ, Spertus JA, Mancini GB, Kostuk W, Chaitman BR, Berman D, Lorin JD, Dada M, Weintraub WS, Boden WE; COURAGE Trial Investigators. Effect of PCI on Long-Term Survival in Patients with Stable Ischemic Heart Disease. N Engl J Med. 2015 Nov 12;373(20):1937-46. doi: 10.1056/NEJMoa1505532. PMID 26559572
- [Derived] Mancini GBJ, Hartigan PM, Shaw LJ, Berman DS, Hayes SW, Bates ER, Maron DJ, Teo K, Sedlis SP, Chaitman BR, Weintraub WS, Spertus JA, Kostuk WJ, Dada M, Booth DC, Boden WE. Predicting outcome in the COURAGE trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation): coronary anatomy versus ischemia. JACC Cardiovasc Interv. 2014 Feb;7(2):195-201. doi: 10.1016/j.jcin.2013.10.017. Epub 2014 Jan 15. PMID 24440015
- [Derived] Mancini GB, Hartigan PM, Bates ER, Chaitman BR, Sedlis SP, Maron DJ, Kostuk WJ, Spertus JA, Teo KK, Dada M, Knudtson M, Berman DS, Booth DC, Boden WE, Weintraub WS. Prognostic importance of coronary anatomy and left ventricular ejection fraction despite optimal therapy: assessment of residual risk in the Clinical Outcomes Utilizing Revascularization and Aggressive DruG Evaluation Trial. Am Heart J. 2013 Sep;166(3):481-7. doi: 10.1016/j.ahj.2013.07.007. Epub 2013 Aug 2. PMID 24016497
- [Derived] Acharjee S, Boden WE, Hartigan PM, Teo KK, Maron DJ, Sedlis SP, Kostuk W, Spertus JA, Dada M, Chaitman BR, Mancini GB, Weintraub WS. Low levels of high-density lipoprotein cholesterol and increased risk of cardiovascular events in stable ischemic heart disease patients: A post-hoc analysis from the COURAGE Trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation). J Am Coll Cardiol. 2013 Nov 12;62(20):1826-33. doi: 10.1016/j.jacc.2013.07.051. Epub 2013 Aug 21. PMID 23973693
- [Derived] Spertus JA, Maron DJ, Cohen DJ, Kolm P, Hartigan P, Weintraub WS, Berman DS, Teo KK, Shaw LJ, Sedlis SP, Knudtson M, Aslan M, Dada M, Boden WE, Mancini GB; Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) Trial Investigators and Coordinators. Frequency, predictors, and consequences of crossing over to revascularization within 12 months of randomization to optimal medical therapy in the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial. Circ Cardiovasc Qual Outcomes. 2013 Jul;6(4):409-18. doi: 10.1161/CIRCOUTCOMES.113.000139. Epub 2013 Jul 9. PMID 23838107
- [Derived] Maron DJ, Hartigan PM, Neff DR, Weintraub WS, Boden WE; COURAGE Trial Investigators. Impact of adding ezetimibe to statin to achieve low-density lipoprotein cholesterol goal (from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation [COURAGE] trial). Am J Cardiol. 2013 Jun 1;111(11):1557-62. doi: 10.1016/j.amjcard.2013.02.005. Epub 2013 Mar 25. PMID 23538020
- [Derived] Farkouh ME, Boden WE, Bittner V, Muratov V, Hartigan P, Ogdie M, Bertolet M, Mathewkutty S, Teo K, Maron DJ, Sethi SS, Domanski M, Frye RL, Fuster V. Risk factor control for coronary artery disease secondary prevention in large randomized trials. J Am Coll Cardiol. 2013 Apr 16;61(15):1607-15. doi: 10.1016/j.jacc.2013.01.044. PMID 23500281
- [Derived] Shaw LJ, Weintraub WS, Maron DJ, Hartigan PM, Hachamovitch R, Min JK, Dada M, Mancini GB, Hayes SW, O'Rourke RA, Spertus JA, Kostuk W, Gosselin G, Chaitman BR, Knudtson M, Friedman J, Slomka P, Germano G, Bates ER, Teo KK, Boden WE, Berman DS. Baseline stress myocardial perfusion imaging results and outcomes in patients with stable ischemic heart disease randomized to optimal medical therapy with or without percutaneous coronary intervention. Am Heart J. 2012 Aug;164(2):243-50. doi: 10.1016/j.ahj.2012.05.018. PMID 22877811
- [Derived] Mancini GB, Hartigan PM, Bates ER, Sedlis SP, Maron DJ, Spertus JA, Berman DS, Kostuk WJ, Shaw LJ, Weintraub WS, Teo KK, Dada M, Chaitman BR, O'Rourke RA, Boden WE; COURAGE Investigators and Coordinators. Angiographic disease progression and residual risk of cardiovascular events while on optimal medical therapy: observations from the COURAGE Trial. Circ Cardiovasc Interv. 2011 Dec 1;4(6):545-52. doi: 10.1161/CIRCINTERVENTIONS.110.960062. Epub 2011 Nov 1. PMID 22045968
- [Derived] Maron DJ, Boden WE, Spertus JA, Hartigan PM, Mancini GB, Sedlis SP, Kostuk WJ, Chaitman BR, Shaw LJ, Berman DS, Dada M, Teo KK, Weintraub WS, O'Rourke RA; COURAGE Trial Research Group. Impact of metabolic syndrome and diabetes on prognosis and outcomes with early percutaneous coronary intervention in the COURAGE (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) trial. J Am Coll Cardiol. 2011 Jul 5;58(2):131-7. doi: 10.1016/j.jacc.2011.02.046. PMID 21718908
- [Derived] Zhang Z, Kolm P, Boden WE, Hartigan PM, Maron DJ, Spertus JA, O'Rourke RA, Shaw LJ, Sedlis SP, Mancini GB, Berman DS, Dada M, Teo KK, Weintraub WS. The cost-effectiveness of percutaneous coronary intervention as a function of angina severity in patients with stable angina. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):172-82. doi: 10.1161/CIRCOUTCOMES.110.940502. Epub 2011 Feb 8. PMID 21304091
- [Derived] Chaitman BR, Hartigan PM, Booth DC, Teo KK, Mancini GB, Kostuk WJ, Spertus JA, Maron DJ, Dada M, O'Rourke RA, Weintraub WS, Berman DS, Shaw LJ, Boden WE; Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial investigators. Do major cardiovascular outcomes in patients with stable ischemic heart disease in the clinical outcomes utilizing revascularization and aggressive drug evaluation trial differ by healthcare system? Circ Cardiovasc Qual Outcomes. 2010 Sep;3(5):476-83. doi: 10.1161/CIRCOUTCOMES.109.901579. Epub 2010 Jul 27. PMID 20664026
- [Derived] Maron DJ, Boden WE, O'Rourke RA, Hartigan PM, Calfas KJ, Mancini GB, Spertus JA, Dada M, Kostuk WJ, Knudtson M, Harris CL, Sedlis SP, Zoble RG, Title LM, Gosselin G, Nawaz S, Gau GT, Blaustein AS, Bates ER, Shaw LJ, Berman DS, Chaitman BR, Weintraub WS, Teo KK; COURAGE Trial Research Group. Intensive multifactorial intervention for stable coronary artery disease: optimal medical therapy in the COURAGE (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) trial. J Am Coll Cardiol. 2010 Mar 30;55(13):1348-58. doi: 10.1016/j.jacc.2009.10.062. PMID 20338496
- [Derived] Weintraub WS, Boden WE, Zhang Z, Kolm P, Zhang Z, Spertus JA, Hartigan P, Veledar E, Jurkovitz C, Bowen J, Maron DJ, O'Rourke R, Dada M, Teo KK, Goeree R, Barnett PG; Department of Veterans Affairs Cooperative Studies Program No. 424 (COURAGE Trial) Investigators and Study Coordinators. Cost-effectiveness of percutaneous coronary intervention in optimally treated stable coronary patients. Circ Cardiovasc Qual Outcomes. 2008 Sep;1(1):12-20. doi: 10.1161/CIRCOUTCOMES.108.798462. PMID 20031783
- [Derived] Teo KK, Sedlis SP, Boden WE, O'Rourke RA, Maron DJ, Hartigan PM, Dada M, Gupta V, Spertus JA, Kostuk WJ, Berman DS, Shaw LJ, Chaitman BR, Mancini GB, Weintraub WS; COURAGE Trial Investigators. Optimal medical therapy with or without percutaneous coronary intervention in older patients with stable coronary disease: a pre-specified subset analysis of the COURAGE (Clinical Outcomes Utilizing Revascularization and Aggressive druG Evaluation) trial. J Am Coll Cardiol. 2009 Sep 29;54(14):1303-8. doi: 10.1016/j.jacc.2009.07.013. PMID 19778673
- [Derived] Weintraub WS, Spertus JA, Kolm P, Maron DJ, Zhang Z, Jurkovitz C, Zhang W, Hartigan PM, Lewis C, Veledar E, Bowen J, Dunbar SB, Deaton C, Kaufman S, O'Rourke RA, Goeree R, Barnett PG, Teo KK, Boden WE; COURAGE Trial Research Group; Mancini GB. Effect of PCI on quality of life in patients with stable coronary disease. N Engl J Med. 2008 Aug 14;359(7):677-87. doi: 10.1056/NEJMoa072771. PMID 18703470
- [Derived] Shaw LJ, Berman DS, Maron DJ, Mancini GB, Hayes SW, Hartigan PM, Weintraub WS, O'Rourke RA, Dada M, Spertus JA, Chaitman BR, Friedman J, Slomka P, Heller GV, Germano G, Gosselin G, Berger P, Kostuk WJ, Schwartz RG, Knudtson M, Veledar E, Bates ER, McCallister B, Teo KK, Boden WE; COURAGE Investigators. Optimal medical therapy with or without percutaneous coronary intervention to reduce ischemic burden: results from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial nuclear substudy. Circulation. 2008 Mar 11;117(10):1283-91. doi: 10.1161/CIRCULATIONAHA.107.743963. Epub 2008 Feb 11. PMID 18268144
- [Derived] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127